CLINICAL TRIAL: NCT02352038
Title: Randomized Controlled Trial of a Novel Laser-aided Orthodontic-periodontal Treatment Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yanqi Yang, Clinical assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HMRF01121056
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Periodontal Disease
Keywords: malocclusion; low-level laser therapy
MeSH Terms: conditions — Periodontal Diseases; Malocclusion | interventions — Low-Level Light Therapy; Orthodontics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LLLT group (Experimental): LLLT group: orthodontic treatment and low-level laser therapy
  Interventions: Device: low-level laser therapy; Other: orthodontic treatment
- control group (Placebo Comparator): Control group: orthodontic treatment and no laser treatment.
  Interventions: Other: orthodontic treatment

INTERVENTIONS:
Device: low-level laser therapy — The test teeth will receive LLLT using a 940 nanometer diode laser (EZLASE; BIOLASE Technology Inc., Irvine, CA, USA) with output power of 330 milliwatt. The experimental side was irradiated for 30 s in two sessions, delivering an energy density of 7 Joules per square centimeter.
  Arms: LLLT group
Other: orthodontic treatment — Orthodontic treatment will be carried out using preadjusted appliances with bonded 0.022×0.028-square inch brackets/buccal tubes and 0.014-inch NiTi archwires as the first archwires. The treatment or the major part of the treatment will be completed in 12 months.

SUMMARY:
The aim of the study is to assess the effects of low-level laser therapy (LLLT) in patients with periodontitis during orthodontic-periodontal treatment for 12 months on the following aspects: (1) Effects on periodontal status; (2) Effects on alveolar bone remodeling; (3) Effects on cervical dentin sensitivity; (4) Effects on pain and quality of life.

To eliminate any bias, the investigators will initially hypothesize that there is no difference in periodontal status, jawbone remodeling, tooth sensitivity, pain and quality of life in patients having teeth with chronic periodontitis and receiving LLLT with orthodontic treatment versus teeth undergoing orthodontic treatment without incorporation of LLLT.

DETAILED DESCRIPTION:
On the basis of the investigators' pilot study results, 35 patients with chronic periodontitis will be recruited and initially treated for inflammation. Using a randomized split-mouth design,the teeth in experimental (laser) group will receive LLLT while the teeth in the control (placebo) group will receive no laser treatment. The effects of LLLT in orthodontic-periodontal treatment on periodontal inflammation control, jawbone remodeling, reduction of tooth sensitivity, pain relief and quality of life will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically health (with special regard to disease affecting tissue repair);
2. No medications required for periodontal therapy and no use of any antibiotic and/or anti-inflammatory medication in the preceding month;
3. Chronic periodontitis with at least two pairs (clinically matched) displaced single-rooted teeth (each pair of teeth is in the same arch but in two contralateral hemi-arches respectively belonging to the same tooth typology) having at least one site probing depth of 5 mm or more, interproximal attachment loss of 3 mm or more, and radiographic signs of alveolar bone loss.
4. Periodontal status confirmed by periodontal evaluation remains stable for at least 6 months after complete periodontal treatment.

Exclusion Criteria:

1. smoking;
2. pregnancy;
3. under orthodontic treatment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
inflammatory cytokine levels in the gingival cervical fluid | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqi Yang, Principal Investigator — The University of Hong Kong
Locations (1):
- The Prince Philip Dental Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of individual participant data has not been decided yet.